CLINICAL TRIAL: NCT06680934
Title: Patient Registry for Individuals With CABP2-Associated Hearing Loss
Brief Title: CABP2 Patient Registry and Natural History Study
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Tobias Moser, Prof., University Medical Center Goettingen
Other Study IDs: 17/8/22 v2.1 - 2023-02528
Record Dates: First submitted 2024-11-03; First posted 2024-11-08 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: CABP2-related Auditory Synaptopathy; Hearing Impairment
Keywords: CABP2 patient registry; Patient registry; DFNB93
MeSH Terms: conditions — Hearing Loss | interventions — Audiometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CABP2 participant group: Individuals with hearing impairment who have a molecular genetic diagnosis involving CABP2
  Interventions: Diagnostic Test: Molecular genetic testing and audiometry

INTERVENTIONS:
Diagnostic Test: Molecular genetic testing and audiometry — Genetic testing and audiometry are the interventions of interest

SUMMARY:
This registry is designed to collect comprehensive information about the molecular genetic diagnoses and clinical information of individuals with CABP2-associated hearing impairment to support a natural history study.

DETAILED DESCRIPTION:
A patient registry, in both German and English languages, has been established for patients with hereditary hearing impairment due to variants in CABP2. The study is conducted in accordance with the current version of the Declaration of Helsinki. The study protocol and database structure have been approved by the Ethics Committee of the University Medical Center Goettingen.

ELIGIBILITY:
Inclusion Criteria:

* A molecular genetic diagnosis involving biallelic variants in CAPB2 and audiometry

Exclusion Criteria:

* Patients with evidence of non-CABP2 molecular genetic diagnoses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with hearing impairment who have a molecular genetic diagnosis involving CABP2
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2049-08-16 (Estimated); Study Completion 2049-08-16 (Estimated)

PRIMARY OUTCOMES:
Pure-tone audiometry | 1 year, year 1, according to participant consent
  Pure tone audiometry is a behavioral hearing test used to measure an individual's hearing threshold levels
Speech audiometry | 1 year, year 1, according to participant consent
  Speech audiometry is a test or series of tests to determine a patient's ability to discriminate speech sounds and hearing speech or speech in noise

SECONDARY OUTCOMES:
Otoacoustic emission thresholds | 1 year, year 1, according to participant consent
  Otoacoustic emission thresholds serve as indicators of integrity and function of the outer hair cells in the cochlea
Auditory brainstem response | 1 year, year 1, according to participant consent
  Auditory brainstem response tests the functional status of the auditory neural pathway

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Moser, MD, Study Director — University Medical Center Goettingen; Bernd Wollnik, MD, Principal Investigator — University Medical Center Goettingen; Nicola Strenzke, MD, Principal Investigator — University Medical Center Goettingen; Barbara Vona, PhD, Principal Investigator — University Medical Center Goettingen
Locations (1):
- University Medical Center Goettingen, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: No
Pseudonymized data will be published in publications

REFERENCES:
- [Result] Vona B, Wollnik B, Strenzke N, Pangrsic T, Moser T. Is CABP2-Associated Hearing Loss (DFNB93) a Gene Therapy Target? Preclinical Progress and Patient Registry. MedComm (2020). 2025 Sep 8;6(9):e70363. doi: 10.1002/mco2.70363. eCollection 2025 Sep. PMID 40927552
- See also: Registry website in English — http://www.auditory-neuroscience.uni-goettingen.de/cabp2_registry_en.html
- See also: Registry website in German — http://www.auditory-neuroscience.uni-goettingen.de/cabp2_registry.html

DOCUMENTS (1):
  • Study Protocol (2025-05-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT06680934/Prot_000.pdf